CLINICAL TRIAL: NCT05096793
Title: Acute Supplementation With Beta-Alanine Improves Performance in Aerobic-anaerobic Transition Zones in Endurance Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Alvaro Huerta Ojeda, Principal Investigator, University of Americas
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 04102021; 04102021 (Other: Uamericas)
Record Dates: First submitted 2021-10-04; First posted 2021-10-27 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Beta-alanine
Keywords: beta-alanine; ergogenic aid; physical performance; aerobic-anaerobic transition zones; maximal aerobic speed
MeSH Terms: interventions — beta-Alanine

STUDY DESIGN:
Intervention Model Description: The experimental design applied was randomized cross-over and double-blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): the distance in the 6-MRT compared to baseline
  Interventions: Dietary Supplement: beta alanine
- Low doses (Experimental): the distance in the 6-MRT compared to baseline
  Interventions: Dietary Supplement: beta alanine
- High doses (Experimental): the distance in the 6-MRT compared to baseline
  Interventions: Dietary Supplement: beta alanine

INTERVENTIONS:
Dietary Supplement: beta alanine — On day 1, all participants completed the 6-MRT corresponding to baseline. Then, on days 2 and 3, each participant performed the 6-MRT with 30 mg·kg-1 and 45 mg·kg-1 of BA (low and high-dose trials, respectively). BA was purchased in powder format from a factory specializing in sports supplements. BA was colorless when diluted in water and had a characteristic taste. This format of BA (powder) allowed personalized dosing for each participant. The research team performed the personalized dosing before the application of the treatment. Between the evaluation days, there was 72 hours difference. The 30 mg·kg-1 or 45 mg·kg-1 BA administration was done with a double-blind method. Thus, on day 2, 50% of the sample performed the 6-MRT supplemented with 30 mg·kg-1 BA, while the other 50% performed the 6-MRT with 45 mg·kg-1 BA. On day 3, those participants who completed the 6-MRT with 30 mg·kg-1 BA now performed with 45 mg·kg-1 BA and vice versa.

SUMMARY:
The use of beta-alanine (BA) to increase physical performance is widely documented. However, the acute effect of this amino acid on maximal tests in the aerobic-anaerobic transition zone is still uncertain. The objective of this study was to determine the acute effect of low and high-dose BA trials on maximal aerobic speed (MAS) in endurance athletes. We hypothesized that high doses of BA have a greater effect than low doses, both compared to baseline. Twelve male endurance athletes volunteered for the study. The experimental design applied was randomized cross-over, double-blind. Treatment included three 6-minute run tests (6-MRT), the first as a baseline, then randomized 6-MRT with low (30 mg·kg-1) and high (45 mg·kg-1) dose BA trials. The 6-MRTs were separated by 72 hours. The main variable of the study was the distance (m) performed in the 6-MRT. Differences between tests were established through ANOVA and Tukey's multiple comparison tests (p < 0.05).

DETAILED DESCRIPTION:
In this original research, we determined the acute effect of low (30 mg·kg-1) and high-dose (45 mg·kg-1) BA trials on maximal aerobic speed (MAS) in endurance athletes. At the same time, we compared the effect size with of BA.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterion was years of training for endurance events (participants had a minimum of two years running middle-distance and long-distance events).

Exclusion Criteria:

* The exclusion criterion was the inability to perform the 6-minute run test

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
6-minute race test (meters) | at the end of the 6 minute test
  The test was performed on an official 400 m athletic track simultaneously every measurement day (09:00 - 11:00 a.m.) and under similar climatic conditions (temperature = 16 - 18° C and relative humidity = 70 - 80%). Also, to simulate the reality of the competition, the 6-MRT was performed in subgroups of three participants. These subgroups were maintained throughout the intervention, modifying only the dose of BA ingested.

SECONDARY OUTCOMES:
Lactate | at the end of the 6 minute test
  A lactometer (h/p/cosmos®) was used to measure capillary [La]. This lactometer generates an enzymatic-amperometric detection of lactate with an accuracy of ± 3% (minimum standard deviation of 0.2 mmol·L-1), sample volume 0.2 μL, and with a measurement range of 0.5-25.0 mmol·L-1.
Heart Rate | at the end of the 6 minute test
  A heart rate monitor (Polar H10®) was used to measure HR, while the data was stored using the Polar Beat® application.

CONTACTS AND LOCATIONS:
Overall Officials: Hernán Cañon, Ph.D., Study Director — University of Americas
Locations (1):
- Uamericas, Viña del Mar, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trexler ET, Smith-Ryan AE, Stout JR, Hoffman JR, Wilborn CD, Sale C, Kreider RB, Jager R, Earnest CP, Bannock L, Campbell B, Kalman D, Ziegenfuss TN, Antonio J. International society of sports nutrition position stand: Beta-Alanine. J Int Soc Sports Nutr. 2015 Jul 15;12:30. doi: 10.1186/s12970-015-0090-y. eCollection 2015. PMID 26175657
- [Result] Boldyrev AA, Aldini G, Derave W. Physiology and pathophysiology of carnosine. Physiol Rev. 2013 Oct;93(4):1803-45. doi: 10.1152/physrev.00039.2012. PMID 24137022
- [Result] Bex T, Chung W, Baguet A, Achten E, Derave W. Exercise training and Beta-alanine-induced muscle carnosine loading. Front Nutr. 2015 May 7;2:13. doi: 10.3389/fnut.2015.00013. eCollection 2015. PMID 25988141
- [Result] Peeling P, Binnie MJ, Goods PSR, Sim M, Burke LM. Evidence-Based Supplements for the Enhancement of Athletic Performance. Int J Sport Nutr Exerc Metab. 2018 Mar 1;28(2):178-187. doi: 10.1123/ijsnem.2017-0343. Epub 2018 Feb 21. PMID 29465269
- [Result] Santesteban Moriones V, Ibanez Santos J. [Ergogenic aids in sport]. Nutr Hosp. 2017 Feb 1;34(1):204-215. doi: 10.20960/nh.997. Spanish. PMID 28244793
- [Result] Mate-Munoz JL, Lougedo JH, Garnacho-Castano MV, Veiga-Herreros P, Lozano-Estevan MDC, Garcia-Fernandez P, de Jesus F, Guodemar-Perez J, San Juan AF, Dominguez R. Effects of beta-alanine supplementation during a 5-week strength training program: a randomized, controlled study. J Int Soc Sports Nutr. 2018 Apr 25;15:19. doi: 10.1186/s12970-018-0224-0. eCollection 2018. PMID 29713250
- [Result] Bassinello D, de Salles Painelli V, Dolan E, Lixandrao M, Cajueiro M, de Capitani M, Saunders B, Sale C, Artioli GG, Gualano B, Roschel H. Beta-alanine supplementation improves isometric, but not isotonic or isokinetic strength endurance in recreationally strength-trained young men. Amino Acids. 2019 Jan;51(1):27-37. doi: 10.1007/s00726-018-2593-8. Epub 2018 Jun 15. PMID 29905904
- [Result] Furst T, Massaro A, Miller C, Williams BT, LaMacchia ZM, Horvath PJ. beta-Alanine supplementation increased physical performance and improved executive function following endurance exercise in middle aged individuals. J Int Soc Sports Nutr. 2018 Jul 11;15(1):32. doi: 10.1186/s12970-018-0238-7. PMID 29996843
- [Result] Santana JO, de Freitas MC, Dos Santos DM, Rossi FE, Lira FS, Rosa-Neto JC, Caperuto EC. Beta-Alanine Supplementation Improved 10-km Running Time Trial in Physically Active Adults. Front Physiol. 2018 Aug 8;9:1105. doi: 10.3389/fphys.2018.01105. eCollection 2018. PMID 30135662
- [Result] Huerta-Ojeda A, Contreras-Montilla O, Galdames-Maliqueo S, Jorquera-Aguilera C, Fuentes-Kloss R, Guisado-Barrilao R. [Effects of acute supplementation with beta-alanine on a limited time test at maximum aerobic speed on endurance athletes]. Nutr Hosp. 2019 Jul 1;36(3):698-705. doi: 10.20960/nh.02310. Spanish. PMID 31144977
- [Result] Kindermann W, Simon G, Keul J. The significance of the aerobic-anaerobic transition for the determination of work load intensities during endurance training. Eur J Appl Physiol Occup Physiol. 1979 Sep;42(1):25-34. doi: 10.1007/BF00421101. PMID 499194
- [Result] Huerta Ojeda A, Tapia Cerda C, Poblete Salvatierra MF, Barahona-Fuentes G, Jorquera Aguilera C. Effects of Beta-Alanine Supplementation on Physical Performance in Aerobic-Anaerobic Transition Zones: A Systematic Review and Meta-Analysis. Nutrients. 2020 Aug 19;12(9):2490. doi: 10.3390/nu12092490. PMID 32824885
- [Result] Poole DC, Jones AM. Measurement of the maximum oxygen uptake V̇o2max: V̇o2peak is no longer acceptable. J Appl Physiol (1985). 2017 Apr 1;122(4):997-1002. doi: 10.1152/japplphysiol.01063.2016. Epub 2017 Feb 2. PMID 28153947
- [Result] Billat LV, Koralsztein JP. Significance of the velocity at VO2max and time to exhaustion at this velocity. Sports Med. 1996 Aug;22(2):90-108. doi: 10.2165/00007256-199622020-00004. PMID 8857705
- [Result] Faude O, Kindermann W, Meyer T. Lactate threshold concepts: how valid are they? Sports Med. 2009;39(6):469-90. doi: 10.2165/00007256-200939060-00003. PMID 19453206
- [Result] Outlaw JJ, Smith-Ryan AE, Buckley AL, Urbina SL, Hayward S, Wingfield HL, Campbell B, Foster C, Taylor LW, Wilborn CD. Effects of beta-Alanine on Body Composition and Performance Measures in Collegiate Women. J Strength Cond Res. 2016 Sep;30(9):2627-37. doi: 10.1519/JSC.0000000000000665. PMID 25486294
- [Result] Stautemas J, Everaert I, Lefevere FBD, Derave W. Pharmacokinetics of beta-Alanine Using Different Dosing Strategies. Front Nutr. 2018 Aug 17;5:70. doi: 10.3389/fnut.2018.00070. eCollection 2018. PMID 30175101
- [Result] Perim P, Marticorena FM, Ribeiro F, Barreto G, Gobbi N, Kerksick C, Dolan E, Saunders B. Can the Skeletal Muscle Carnosine Response to Beta-Alanine Supplementation Be Optimized? Front Nutr. 2019 Aug 27;6:135. doi: 10.3389/fnut.2019.00135. eCollection 2019. PMID 31508423
- [Result] Harriss DJ, MacSween A, Atkinson G. Ethical Standards in Sport and Exercise Science Research: 2020 Update. Int J Sports Med. 2019 Dec;40(13):813-817. doi: 10.1055/a-1015-3123. Epub 2019 Oct 15. No abstract available. PMID 31614381
- [Result] Cooper KH. A means of assessing maximal oxygen intake. Correlation between field and treadmill testing. JAMA. 1968 Jan 15;203(3):201-4. No abstract available. PMID 5694044
- [Result] Ojeda AH, Barahona-Fuentes G, Maliqueo SG. A qualitative scale of the 6-minute race test to evaluate maximum aerobic speed in physically active people from 18 to 25 years. J Phys Ther Sci. 2021 Apr;33(4):316-321. doi: 10.1589/jpts.33.316. Epub 2021 Apr 6. PMID 33935354
- [Result] Hopkins WG, Marshall SW, Batterham AM, Hanin J. Progressive statistics for studies in sports medicine and exercise science. Med Sci Sports Exerc. 2009 Jan;41(1):3-13. doi: 10.1249/MSS.0b013e31818cb278. PMID 19092709
- [Result] Tanokura M, Tasumi M, Miyazawa T. 1H nuclear magnetic resonance studies of histidine-containing di- and tripeptides. Estimation of the effects of charged groups on the pKa value of the imidazole ring. Biopolymers. 1976 Feb;15(2):393-401. doi: 10.1002/bip.1976.360150215. No abstract available. PMID 2351
- [Result] Suzuki Y, Nakao T, Maemura H, Sato M, Kamahara K, Morimatsu F, Takamatsu K. Carnosine and anserine ingestion enhances contribution of nonbicarbonate buffering. Med Sci Sports Exerc. 2006 Feb;38(2):334-8. doi: 10.1249/01.mss.0000185108.63028.04. PMID 16531904
- [Result] Hill CA, Harris RC, Kim HJ, Harris BD, Sale C, Boobis LH, Kim CK, Wise JA. Influence of beta-alanine supplementation on skeletal muscle carnosine concentrations and high intensity cycling capacity. Amino Acids. 2007 Feb;32(2):225-33. doi: 10.1007/s00726-006-0364-4. Epub 2006 Jul 28. PMID 16868650
- [Result] Artioli GG, Gualano B, Smith A, Stout J, Lancha AH Jr. Role of beta-alanine supplementation on muscle carnosine and exercise performance. Med Sci Sports Exerc. 2010 Jun;42(6):1162-73. doi: 10.1249/MSS.0b013e3181c74e38. PMID 20479615
- [Result] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Result] Decombaz J, Beaumont M, Vuichoud J, Bouisset F, Stellingwerff T. Effect of slow-release beta-alanine tablets on absorption kinetics and paresthesia. Amino Acids. 2012 Jul;43(1):67-76. doi: 10.1007/s00726-011-1169-7. Epub 2011 Dec 3. PMID 22139410